CLINICAL TRIAL: NCT04101110
Title: Epidemiology, Risk Factors and Outcomes of Transition of Acute Kidney Injury to Chronic Kidney Disease in Critically Ill Patients
Brief Title: Transition of Acute Kidney Injury to Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa A Mohammed, Prinsipal Investigator, Assiut University
Other Study IDs: EROT
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2020-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Renal biopsy — Kidney biopsy will be done to understand the nature and degree of structural kidney damage

SUMMARY:
Acute kidney injury is a complex clinical syndrome,associated with high short and long- term morbidity and mortality in critical ill patients.Acute kidney injury outcomes may vary from a complete resolution to a partial or incomplete recovery of renal function leading to increased mortality,prolonged hospitalization and risk of chronic comorbidities .

The precise mechanism of acute kidney injury to chronic kidney disease transition is complex and not completely understood,especially in humans .Acute kidney injury outcomes depend upon the balance of adaptive and maladaptive repair.

DETAILED DESCRIPTION:
Acute kidney injury is a life threatening and disabling complication of critical illness encountered in 25 -50%h of intensive care unit admission.Acute kidney injury is a complex clinical syndrome,associated with high short and long- term morbidity and mortality in critical ill patients.

Acute kidney injury outcomes may vary from a complete resolution to a partial or incomplete recovery of renal function leading to increased mortality,prolonged hospitalization and risk of chronic comorbidities like cardiovascular disease,chronic kidney disease and subsequent progression to end stage renal disease.Several studies have suggested a causal link between acute kidney injury and the consequent development of chronic kidney disease.the severity,frequency and duration of acute kidney injury are key factors in this process.

The precise mechanism of transition of acute kidney injury to chronic kidney disease is complex and not completely understood,especially in humans and several pathways have been proposed. Different animal studies have used ischemia-reperfusion and nephrotoxic injuries to investigate the pathophysiologic event involved in acute kidney injury to chronic kidney disease transition ,mainly focusing in the development of specific histological changes .Acute kidney injury outcomes depend, at the tissue level,upon the balance of adaptive and maladaptive repair. An adaptive response to injury usually leads to renal recovery with a complete resolution of pathological changes during acute kidney injury episode(resolution of inflammatory cell infiltration, regeneration of tubular cells,decrease in biomarkers of injury )without long term consequences .However,severe and repeated injury can result in a maladaptive repair,characterized by a permanent reduction in kidney function associated with significant structural changes (persistent expression of pro-fibrotic factors and development of interstitial fibrosis, delayed resolution of inflammation,permanent cell cycle arrest of tubular cells, microvascular rarefaction,renin angiotensin system activation).

The incidence rate of renal progression following acute kidney injury has been estimated to be 4.9 events /100 patient-year and is particularly increase in elderly.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥18 years;
* patients suffering an acute kidney injury (defined by Acute kidney injury network (AKIN) score ≥1)during ICU stay.

Exclusion Criteria:

* patients <18 years;
* pregnant woman;
* End stage renal disease (ESRD)prior to ICU admission;
* Refusal to participate in the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients attending Assiut university hospitals critical care unit and developing acute kidney injury during their stay.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic kidney disease | Baseline
  Incidence of chronic kidney disease defined by a decreased glomerular filtration rate under 60 mL/minute/1.73m2

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sileanu FE, Murugan R, Lucko N, Clermont G, Kane-Gill SL, Handler SM, Kellum JA. AKI in low-risk versus high-risk patients in intensive care. Clin J Am Soc Nephrol. 2015 Feb 6;10(2):187-96. doi: 10.2215/CJN.03200314. Epub 2014 Nov 25. PMID 25424992
- [Result] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Result] Singbartl K, Kellum JA. AKI in the ICU: definition, epidemiology, risk stratification, and outcomes. Kidney Int. 2012 May;81(9):819-25. doi: 10.1038/ki.2011.339. Epub 2011 Oct 5. PMID 21975865
- [Result] Goldstein SL, Chawla L, Ronco C, Kellum JA. Renal recovery. Crit Care. 2014 Jan 6;18(1):301. doi: 10.1186/cc13180. PMID 24393370